CLINICAL TRIAL: NCT05826184
Title: Time Restricted Eating With or Without a Fiber Supplement for Weight Management in Pediatric Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Kelsey Nicole Dipman Gabel, Clinial Assistant Professor and Postdoctoral Researcher, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY2022-0745
Record Dates: First submitted 2023-04-10; First posted 2023-04-24 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-02

CONDITIONS: Weight, Body
MeSH Terms: conditions — Body Weight | interventions — Prebiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Time restricted eating (Experimental): Individuals will eat between 12-8pm ad libitum, fasting from 8-12pm.
  Interventions: Behavioral: Time restircted eating
- TRE+ prebiotic supplement (Experimental): Individuals will eat between 12-8pm ad libitum, fasting from 8-12pn with the addition of a prebiotic fiber supplement with the first eating bout of the day.
  Interventions: Behavioral: Time restricted eating + prebiotic

INTERVENTIONS:
Behavioral: Time restircted eating — 8 hour time restricted eating alone
  Arms: Time restricted eating
Behavioral: Time restricted eating + prebiotic — 8 hour TRE with a prebiotic supplement
  Arms: TRE+ prebiotic supplement

SUMMARY:
This study aims to address a critical gap in pediatric oncology survivorship care by exploring innovative solutions to addressing obesity and its comorbidities in pediatric cancer survivors. The majority (99%) of pediatric cancer survivors will develop severe chronic health conditions by age 50, with 96% developing at least one severe/disabling, life threating or fatal chronic health condition. Obesity, cardiovascular, and metabolic diseases are the most common treatment-related late effects among pediatric cancer survivors. Improving diet and reducing obesity has the potential to dramatically improve the quality of life and long-term health of pediatric cancer survivors. Utilization of a prebiotic fiber supplement along with TRE amy improve the gut microbiome, short-chain fatty acid synthesis, and hunger hormones to further improve weight loss with TRE and a greater decrease in cardiometabolic risk. The aims of this study are to test the safety, feasibility, and acceptability of 8-h TRE or 8-h TRE with a fiber supplement among young adult (YA) pediatric cancer survivors. The investigators further strive to examine the preliminary efficacy of TRE on body weight, body composition, glucose regulation, and cardiovascular risk markers. Data obtained will be used to inform a larger efficacy trial of TRE among adolescent and young adult pediatric cancer survivors. Given that a majority of pediatric cancer survivors will develop severe chronic health conditions by age 50, with 96% developing at least one severe/disabling, life threating or fatal chronic health condition exploring accessible nutritional strategies to improve long term health trajectory of 70,000+ AYA diagnosed with cancer each year in the United States. This study of TRE will provide important preliminary evidence of the benefits of this nutrition therapy for YA pediatric cancer survivors. The long-term goal of this line of inquiry is to improve both short and long-term outcomes for YA pediatric cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-39 years old at time of consent
* Completed anti-tumor treatment for pediatric cancer
* BMI 25-39.99 kg/m2
* Able to provide (self or guardian) written informed consent and HIPAA authorization for release of personal health information, via an approved UIC Institutional Review Board (IRB) informed consent form and HIPAA authorization.
* As determined at the discretion of the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

Subjects meeting any of the criteria below may not participate in the study:

* Individuals <18 or >39 years of age
* Individuals on glucoregulatory medication
* Individuals with BMI ≥ 40kg/m2 and < 25kg/m2
* Individuals who are pregnant, trying to become pregnant or breast feeding. A negative serum or urine pregnancy test is required per institutional practice guidelines at screening as well as prior to all DXA scans.
* Shift workers who maintain a work schedule that crosses 12:00 am > 1 day per week
* Individuals with a history of eating disorders
* Active infection requiring systemic therapy
* Uncontrolled HIV/AIDS or active viral hepatitis
* Any mental or medical condition that prevents the patient from giving informed consent or participating in the trial.
* Other major comorbidity, as determined by study PI
* Illicit drug use (excluding self-reported marijuana) or excessive use of alcohol (i.e., > 2 drinks/day)
* Currently participating in Weight Watcher's or another weight loss program with a ≥ 3% weight loss in three months prior to recruitment
* History of: Myocardial infarction, Stroke, Congestive heart failure, Chronic hepatitis, Cirrhosis, Chronic pancreatitis
* History of solid organ transplantation
* Individual does not have access to the Internet
* Individuals who have taken antibiotics < 2 months prior to the initiation of the study
* Individuals who regularly use (≥ 3 times per week) prebiotics, probiotics, synbiotics, prebiotic supplements or laxatives within the past month

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
feasibility of TRE in pediatric cancer survivors | 1 year
  Clinicians will refer ≥ 75% of AYA pediatric cancer survivors that are eligible, we will screen and enroll ≥ 50% of those referred, participants will complete ≥ 80% of planned study visits, and we will retain ≥ 80% of participants in both study arms through the end of the intervention.
acceptance of TRE in pediatric cancer survivors | 12 weeks
  TRE will be acceptable (≥ 16 on acceptability on Diet Satistfaction questionnaire).
Adherence to TRE | 12 weeks
  Adherence to TRE will be ≥ 80% throughout the intervention among participants randomized to this study arm

SECONDARY OUTCOMES:
body weight (kg) | change from week 1-12
  Body weight assessed to the nearest 0.25 kg every week without shoes and in light clothing using a balance beam scale (HealthOMeter, Boca Raton, FL).
Body composition | change from week 1-12
  fat free mass and fat mass via DXA
fasting Insulin | change from week 1-12
  measured by enzymatic kit (uIU/ml)^4
fasting glucose | change from week 1-12
  measured by enzymatic kit (mg/dl)
insulin resistance change | change from week 1-12
  fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5.
Hemoglobin A1c concentration | change from week 1-12
  measured by enzymatic kit
Blood pressure | change from week 1-12
  systolic and diastolic blood pressure with cuff
Heart rate | change from week 1-12
  Heart rate measured by blood pressure cuff
Lipid concentration | change from week 1-12
  measured by enzymatic kit
Gut microbial composition | Change from week 1-12
  16s RNA stool swab
Glucagon like peptide 1 concentration | change from week 1-12
  measured by enzymatic kit
peptide yy concentration | change from week 1-12
  measured by enzymatic kit
circulating short chain fatty acid concentration | change from week 1-12
  measured by enzymatic kit
c-reactive protein concentration | change from week 1-12
  measured by enzymatic kit

OTHER OUTCOMES:
peripheral blood mononuclear cell (PBMC) telomerase activity | change from week 1-12
  measured by enzymatic kit

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey Gabel, PhD, Principal Investigator — UIC
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No